CLINICAL TRIAL: NCT03548220
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of AG-348 in Not Regularly Transfused Adult Subjects With Pyruvate Kinase Deficiency
Brief Title: A Study to Evaluate Efficacy and Safety of AG-348 in Not Regularly Transfused Adult Participants With Pyruvate Kinase Deficiency (PKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG348-C-006
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Pyruvate Kinase Deficiency; Anemia, Hemolytic
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic | interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received a matching placebo to AG-348 tablets, for a period of 12 weeks as an optimized dose. This was followed by matching placebo further, for a period of 12 weeks as a fixed-dose.
  Interventions: Drug: Placebo
- AG-348, 5 mg (Experimental): Participants received AG-348 tablets, 5 milligrams (mg) twice daily (BID), administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
  Interventions: Drug: AG-348
- AG-348, 20 mg (Experimental): Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 20 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
  Interventions: Drug: AG-348
- AG-348, 50 mg (Experimental): Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 50 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: Placebo — Placebo matching AG-348 tablets, administered to maintain the blind.
  Arms: Placebo
Drug: AG-348 — AG-348 tablets.
  Arms: AG-348, 20 mg; AG-348, 5 mg; AG-348, 50 mg

SUMMARY:
Study AG348-C-006 evaluated the efficacy and safety of orally administered AG-348 as compared with placebo in participants with pyruvate kinase (PK) deficiency, who were not regularly receiving blood transfusions. Participants were randomized 1:1 to receive either AG-348 or a matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* Male or female, aged 18 years or older;
* Documented clinical laboratory confirmation of pyruvate kinase (PK) deficiency, defined as documented presence of at least 2 mutant alleles in the PKLR gene, of which at least 1 is a missense mutation;
* Hemoglobin (Hb) concentration less than or equal to 10.0 grams per deciliter (g/dL) regardless of gender (average of at least 2 Hb measurements [separated by a minimum of 7 days] during the Screening Period)
* Considered not regularly transfused, defined as having had no more than 4 transfusion episodes in the 12-month period up to the first day of study treatment and no transfusions in the 3 months prior to the first day of study treatment;
* Received at least 0.8 mg oral folic acid daily for at least 21 days prior to the first dose of study treatment, to be continued daily during study participation.
* Adequate organ function;
* Women of reproductive potential, have a negative serum pregnancy test;
* For women of reproductive potential as well as men with partners who are women of reproductive potential, be abstinent as part of their usual lifestyle, or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of giving informed consent, during the study, and for 28 days following the last dose of study treatment for women and 90 days for men following the last dose of study treatment;
* Willing to comply with all study procedures for the duration of the study;

Exclusion Criteria:

* Homozygous for the R479H mutation or have 2 non-missense mutations, without the presence of another missense mutation, in the PKLR gene;
* Significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data;
* Splenectomy scheduled during the study treatment period or have undergone splenectomy within 12 months prior to signing informed consent;
* Currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo. Prior and subsequent participation in the PK Deficiency Natural History Study (NHS) (NCT02053480) or PK Deficiency Registry is permitted however, concurrent participation is not; participants enrolling in this current study will be expected to temporarily suspend participation in the NHS or Registry;
* Exposure to any investigational drug, device, or procedure within 3 months prior to the first dose of study treatment;
* Prior treatment with a pyruvate kinase activator;
* Prior bone marrow or stem cell transplant;
* Currently pregnant or breastfeeding;
* History of major surgery within 6 months of signing informed consent;
* Currently receiving medications that are strong inhibitors of cytochrome P450 (CYP)3A4, strong inducers of CYP3A4, strong inhibitors of P-glycoprotein (P-gp), or digoxin (a P-gp sensitive substrate medication) that have not been stopped for a duration of at least 5 days or a timeframe equivalent to 5 half-lives (whichever is longer) prior to the first dose of study treatment;
* Currently receiving hematopoietic stimulating agents that have not been stopped for a duration of at least 28 days prior to the first dose of study treatment;
* History of allergy to sulfonamides if characterized by acute hemolytic anemia, drug induced liver injury, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson syndrome, cholestatic hepatitis, or other serious clinical manifestations;
* History of allergy to AG-348 or its excipients;
* Currently receiving anabolic steroids, including testosterone preparations, within 28 days prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (46):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Emory University, Atlanta, Georgia
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Children's Hospital Corporation d/b/a Boston's Children Hospital, Boston, Massachusetts
  - Wayne State University School of Medicine, Children's Hospital of Michigan, Detroit, Michigan
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Houston Methodist Research Institute, Houston, Texas
  - Primary Children's Hospital Univ. of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Hospital Central da Faculdade de Medicina USP Cidade Universitaria, São Paulo, Brazil
- Canada (2):
  - McMaster University - Health Sciences Centre, Hamilton
  - Toronto General Hospital, University Health Network, Toronto
- Institute of Hematology and Blood Transfusion, Prague, Czechia
- University of Copenhagen, Herlev Hospital, Herlev, Denmark
- France (5):
  - CHU Amiens Picardie, Amiens
  - Hopital Saint-Andre, Bordeaux
  - Hôpital Henri-Mondor, Créteil
  - Hôpital de la Timone, Marseille
  - Institut Claudius Regaud, Toulouse
- Germany (2):
  - Charite University Medicine, Berlin
  - Universitätsklinikum Würzburg, Würzburg
- Italy (3):
  - Ospedale Galliera, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - AOU Policlinico, Università della Campania "Luigi Vanvitelli", Napoli
- Japan (6):
  - Tohoku University Hospital, Sendai, Miyagi
  - Kyoto Katsura Hospital, Kyoto
  - Agios Investigative Site, Mie
  - Osaka City General Hospital, Osaka
  - Kansai Medical University, Department of Pediatrics, Hirakata Hospital, Osaka
  - Toho University Omori Medical Center, Tokyo
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Yeungnam University Hospital, Daegu 705-703, South Korea
- Spain (3):
  - Hospital U. Vall d'Hebron Servicio de Hematología Clínica, Barcelona
  - Hospital Clinico Universitario Virgen de la Arricaxa, El Palmar
  - Hospital Universitario La Paz, Madrid
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
- Department of Paediatrics and Thalassaemia Center, Faculty of Medicine Siriraj, Bangkok, Thailand
- Hacettepe University, Ankara, Turkey (Türkiye)
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge
  - The Royal Liverpool and Broadgreen University, Liverpool
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Beers EJ, Al-Samkari H, Grace RF, Barcellini W, Glenthoj A, DiBacco M, Wind-Rotolo M, Xu R, Beynon V, Patel P, Porter JB, Kuo KHM. Mitapivat improves ineffective erythropoiesis and iron overload in adult patients with pyruvate kinase deficiency. Blood Adv. 2024 May 28;8(10):2433-2441. doi: 10.1182/bloodadvances.2023011743. PMID 38330179
- [Derived] Andrae DA, Grace RF, Jewett A, Foster B, Klaassen RJ, Salek S, Li J, Tai F, Boscoe AN, Zagadailov E. Psychometric validation of the Pyruvate Kinase Deficiency Diary and Pyruvate Kinase Deficiency Impact Assessment in adults in the phase 3 ACTIVATE trial. J Patient Rep Outcomes. 2023 Nov 9;7(1):112. doi: 10.1186/s41687-023-00650-3. PMID 37943362
- [Derived] Al-Samkari H, Grace RF, Glenthoj A, Andres O, Barcellini W, Galacteros F, Kuo KHM, Layton DM, Morado Arias M, Viprakasit V, Dong Y, Tai F, Hawkins P, Gheuens S, Morales-Arias J, Gilroy KS, Porter JB, van Beers EJ. Early-onset reduced bone mineral density in patients with pyruvate kinase deficiency. Am J Hematol. 2023 Mar;98(3):E57-E60. doi: 10.1002/ajh.26830. Epub 2023 Jan 9. No abstract available. PMID 36594181
- [Derived] Al-Samkari H, Galacteros F, Glenthoj A, Rothman JA, Andres O, Grace RF, Morado-Arias M, Layton DM, Onodera K, Verhovsek M, Barcellini W, Chonat S, Judge MP, Zagadailov E, Xu R, Hawkins P, Beynon V, Gheuens S, van Beers EJ; ACTIVATE Investigators. Mitapivat versus Placebo for Pyruvate Kinase Deficiency. N Engl J Med. 2022 Apr 14;386(15):1432-1442. doi: 10.1056/NEJMoa2116634. PMID 35417638
- [Derived] Rab MAE, Van Oirschot BA, Kosinski PA, Hixon J, Johnson K, Chubukov V, Dang L, Pasterkamp G, Van Straaten S, Van Solinge WW, Van Beers EJ, Kung C, Van Wijk R. AG-348 (Mitapivat), an allosteric activator of red blood cell pyruvate kinase, increases enzymatic activity, protein stability, and ATP levels over a broad range of PKLR genotypes. Haematologica. 2021 Jan 1;106(1):238-249. doi: 10.3324/haematol.2019.238865. PMID 31974203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were randomized in the study, which was conducted across multiple sites in 14 countries: Brazil, Canada, Denmark, France, Germany, Italy, Japan, Republic of Korea, Netherlands, Spain, Switzerland, Turkey, United Kingdom, and United States. The study was conducted from 9 August 2018 to 9 October 2020.
Pre-assignment Details: Screening was done for a period of 42 days after the participant provided the informed consent. Investigators determined if the participants met all the inclusion criteria and none of the exclusion criteria to receive AG-348 or placebo to determine the optimized dose to be received for 12 weeks as fixed-dose.
Groups:
- Placebo Comparator: Placebo: Participants received a matching placebo to AG-348 tablets, for a period of 12 weeks as an optimized dose. This was followed by matching placebo further, for a period of 12 weeks as a fixed-dose.
- Experimental: AG-348 5 mg: Participants received AG-348 tablets, 5 milligrams (mg) twice daily (BID), administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
- Experimental: AG-348, 20 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 20 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
- Experimental: AG-348, 50 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 50 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
Period: Overall Study
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348 5 mg | Experimental: AG-348, 20 mg | Experimental: AG-348, 50 mg
Started | 40 | 2 | 3 | 35
Completed | 39 | 2 | 3 | 35
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomized.
Groups:
- Experimental: AG-348, 5 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348, 5 mg | Experimental: AG-348, 20 mg | Experimental: AG-348, 50 mg | Total
Number analyzed (Participants) | 40 | 2 | 3 | 35 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (15.92) | 21.5 (4.95) | 48.0 (26.21) | 35.8 (14.07) | 36.6 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 0 | 2 | 22 | 48
  Male | 16 | 2 | 1 | 13 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 34 | 1 | 2 | 25 | 62
  Unknown or Not Reported | 5 | 1 | 1 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 32 | 2 | 3 | 23 | 60
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 0 | 0 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Hemoglobin (Hb) Response (HR)
Description: Hemoglobin response (HR) is defined as a ≥1.5 g/dL (0.93 mmol/L) increase in Hb concentration from baseline that is sustained at 2 or more scheduled assessments at Weeks 16, 20, and 24. The baseline Hb concentration is the average of all available Hb concentrations for a participant during the Screening Period up to the first dose of study treatment. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: Full analysis set included all participants who were randomized.
Measure: Number; unit: percentage of participants
Groups:
- Placebo Comparator: Placebo: Participants received matching placebo to AG-348 tablets, for a period of 12 weeks as an optimized dose. This was followed by matching placebo further, for a period of 12 weeks as a fixed-dose.
- Experimental: AG-348: Participants received AG-348 tablets, 5 mg for 4 weeks followed by the respective optimized dose of 5 mg or 20 mg or 50 mg BID as determined by the investigator, administered orally, up to Weeks 8 and 12 respectively, as an optimized dose and continued to receive the same dose for a period of 12 weeks as a fixed-dose.
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 40 | 40
percentage of participants | 0 | 40.0
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p < 0.0001, Exact Cochran-Mantel-Haenszel — 2-sided p-value

2. Secondary Outcome: Average Change From Baseline in Hb Concentration at Weeks 16, 20 and 24
Description: This is the change in Hb concentration at Weeks 16, 20 and 24 compared to baseline. Data presented represents the value of the change from baseline averaged over Weeks 16, 20 and 24. Baseline was defined as the average of all screening assessments within 45 (42+3) days before randomization for participants randomized and not dosed or before start of study treatment for participants randomized and dosed. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: Full analysis set included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: grams per liter (g/L)
Groups:
- Placebo Comparator: Placebo: Participants received matching placebo to AG-348 tablets, for a period of 12 weeks as an optimized dose. This was followed by matching placebo further, for a period of 12 weeks as a fixed dose.
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 40 | 40
grams per liter (g/L) | -1.48 (2.082) | 16.73 (2.075)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measure; LS Mean Difference = 18.21, 95% CI 2-sided [12.41 to 24.01] — Standard error = 2.913

3. Secondary Outcome: Maximum Change From Baseline in Hb Concentration
Description: This is the maximum change from baseline in Hb concentration up to Week 24. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, up to Week 24
Population: Full analysis set included all participants who were randomized. Overall number of participants analyzed is the number of participants evaluated for the outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 39 | 39
g/L | 4.76 (4.217) | 23.94 (21.367)

4. Secondary Outcome: Time to Achieve an Increase in Hb Concentration of 1.5 g/dL or More
Description: This is the time taken to first achieve an increase of hemoglobin concentration of 1.5 g/dL or more from baseline. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, up to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 0 | 17
weeks |  | 7.66 (4.050)

5. Secondary Outcome: Average Change From Baseline in Indirect Bilirubin at Weeks 16, 20 and 24
Description: The change from baseline in indirect bilirubin levels was summarized. Indirect bilirubin is a marker for hemolysis. Data presented represents the value of the change from baseline averaged over Weeks 16, 20 and 24. Baseline was defined as the average of all screening assessments within 45 (42+3) days before randomization for participants randomized and not dosed or before the start of study treatment for participants randomized and dosed. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: micromoles per liter (μmol/L)
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 39 | 37
micromoles per liter (μmol/L) | 5.10 (4.061) | -21.16 (4.228)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measure; LS Mean Difference = -26.26, 95% CI 2-sided [-37.82 to -14.70] — Standard error = 5.788

6. Secondary Outcome: Average Change From Baseline in Lactic Acid Dehydrogenase (LDH) at Weeks 16, 20 and 24
Description: The change from baseline in LDH levels was summarized. LDH is a marker for hemolysis. Data presented represents the value of the change from baseline averaged over Weeks 16, 20 and 24. Baseline was defined as the average of all screening assessments within 45 (42+3) days before randomization for participants randomized and not dosed or before the start of study treatment for participants randomized and dosed. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units per litre (U/L)
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 40 | 39
units per litre (U/L) | -21.18 (16.040) | -91.99 (16.222)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p = 0.0027, Mixed-effect Model Repeated Measure; LS Mean Difference = -70.81, 95% CI 2-sided [-115.88 to -25.74] — Standard error = 22.488

7. Secondary Outcome: Average Change From Baseline in Haptoglobin at Weeks 16, 20 and 24
Description: The change from baseline in haptoglobin levels was summarized. Haptoglobin levels are markers for hemolysis. Data presented represents the value of the change from baseline averaged over Weeks 16, 20 and 24. Baseline was defined as the average of all screening assessments within 45 (42+3) days before randomization for participants randomized and not dosed or before the start of study treatment for participants randomized and dosed. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: Full analysis set included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 40 | 40
g/L | 0.012 (0.0412) | 0.169 (0.0408)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p = 0.0079, Mixed-effect Model Repeated Measure; LS Mean Difference = 0.158, 95% CI 2-sided [0.043 to 0.273] — Standard error = 0.0578

8. Secondary Outcome: Average Change From Baseline in Reticulocyte Percentages at Weeks 16, 20 and 24
Description: The change from baseline in reticulocyte percentage was summarized. Reticulocyte levels are markers for hematopoietic activity. Data presented represents the value of the change from baseline averaged over Weeks 16, 20 and 24. Baseline was defined as the average of all screening assessments within 45 (42+3) days before randomization for participants randomized and not dosed or before the start of study treatment for participants randomized and dosed. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Weeks 16, 20, 24
Population: Full analysis set included all participants who were randomized.
Measure: Least Squares Mean (Standard Error); unit: Reticulocyte percentages
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 40 | 40
Reticulocyte percentages | 0.0038 (0.01390) | -0.0973 (0.01401)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeated Measure; LS Mean Difference = -0.1011, 95% CI 2-sided [-0.1391 to -0.0632] — Standard error = 0.01904

9. Secondary Outcome: Change From Baseline in Pyruvate Kinase Deficiency Diary (PKDD) Score at Week 24
Description: The PKDD is a 7-item patient reported outcome (PRO) measure of the core signs and symptoms associated with PK deficiency in adults. Participants rate their experience with symptoms of PK deficiency on the present day. The symptoms include those associated with tiredness, jaundice, bone pain, shortness of breath, and energy level. The score ranges from 25 to 76, with higher scores indicating a higher disease burden. The change from baseline in PKDD weekly scores was evaluated. A negative change from baseline indicates a lower disease burden. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 36 | 37
score on a scale | -2.05 (0.976) | -5.16 (0.955)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p = 0.0247, Mixed-effect Model Repeated Measure; LS Mean Difference = -3.11, 95% CI 2-sided [-5.80 to -0.41] — Standard error = 1.352

10. Secondary Outcome: Change From Baseline in Pyruvate Kinase Deficiency Impact Assessment (PKDIA) Score at Week 24
Description: The PKDIA is a 12-item patient reported outcome (PRO) measure of the common impacts of PK deficiency on activities of daily living. Participants rate how PK deficiency has impacted aspects of daily living in the past 7 days, including impacts on relationships; perceived appearance; work performance; and leisure, social, mental, and physical activities. The score range is 30 to 76, with higher scores indicating a higher disease burden. The change from baseline in PKDIA scores was evaluated. A negative change from baseline indicates a lower disease burden. As pre-specified in the protocol, the data for this outcome measure is summarized between the active arm vs the placebo arm (AG-348 5 mg, 20 mg and 50 mg arms are analyzed and reported together in comparison to Placebo).
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348
Number analyzed (Participants) | 39 | 39
score on a scale | -1.39 (1.157) | -4.65 (1.123)
Statistical Analysis 1: Comparison: Placebo Comparator: Placebo vs Experimental: AG-348; Test type: Superiority; p = 0.0421, Mixed-effect Model Repeated Measure; LS Mean Difference = -3.25, 95% CI 2-sided [-6.39 to -0.12] — Standard error = 1.574

11. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From signing of informed consent form to the end of study, including follow-up (up to Day 197)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Groups:
- Experimental: AG-348 5 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose
- Experimental: AG-348 20 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 20 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
- Experimental: AG-348 50 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 50 mg BID at Week 12, and participants then received that optimized dose for a period of 12 weeks as a fixed dose.
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348 5 mg | Experimental: AG-348 20 mg | Experimental: AG-348 50 mg
Number analyzed (Participants) | 39 | 2 | 3 | 35
percentage of participants | 89.7 | 50.0 | 100 | 88.6

12. Secondary Outcome: Area Under the Curve From Time 0 to the Last Quantifiable Concentration [AUC(0-last)] for AG-348 at Week 12
Time Frame: Pre-dose, 30 minutes and 1, 2, 4 and 8 hours post-dose on Day 85 (Week 12)
Population: Pharmacokinetic analysis population consisted of all participants who were enrolled and received a dose of study medication (mitapivat) with at least 1 non-zero pharmacokinetic plasma concentration of mitapivat at the Week 12 visit. Overall number of participants analyzed is the number of participants evaluated for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- AG-348, 5mg: Participants received 5mg AG-348 tablets BID at Week 12.
- AG-348, 20 mg: Participants received 20mg AG-348 tablets BID at Week 12.
- AG-348, 50mg: Participants received 50mg AG-348 tablets BID at Week 12.
Arm/Group | AG-348, 5mg | AG-348, 20 mg | AG-348, 50mg
Number analyzed (Participants) | 2 | 3 | 24
h*ng/mL | 565.9 (NA) — Data was not reported due to small size of sample. | 1481.2 (26.9) | 2973.3 (35.6)

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) for AG-348
Time Frame: Pre-dose, 30 minutes and 1, 2, 4 and 8 hours post-dose on Day 85 (Week 12)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | AG-348, 5mg | AG-348, 20 mg | AG-348, 50mg
Number analyzed (Participants) | 2 | 3 | 26
Nanograms per milliliter (ng/mL) | 156.9 (NA) — Data not reported due to small size of sample. | 373.1 (13.6) | 1033 (31.2)

14. Secondary Outcome: Time to Cmax (Tmax) for AG-348
Time Frame: Pre-dose, 30 minutes and 1, 2, 4 and 8 hours post-dose on Day 85 (Week 12)
Population: as for outcome 12
Measure: Median (Full Range); unit: hours (h)
Groups:
- AG-348, 20mg: Participants received 20mg AG-348 tablets BID at Week 12.
Arm/Group | AG-348, 5mg | AG-348, 20mg | AG-348, 50mg
Number analyzed (Participants) | 2 | 3 | 26
hours (h) | 0.75 [0.50 to 1.00] | 1.02 [0.92 to 2.17] | 0.50 [0.42 to 1.92]

15. Secondary Outcome: Time to Last Measurable Concentration (Tlast) for AG-348
Time Frame: Pre-dose, 30 minutes and 1, 2, 4 and 8 hours post-dose on Day 85 (Week 12)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Groups:
- AG-346, 50mg: Participants received 50mg AG-348 tablets BID at Week 12.
Arm/Group | AG-348, 5mg | AG-348, 20mg | AG-346, 50mg
Number analyzed (Participants) | 2 | 3 | 24
hours (h) | 7.787 (NA) — Data not reported due to small size of sample. | 7.809 (4.2) | 7.162 (28.0)

16. Secondary Outcome: Exposure-Response Relationship of Adverse Event (Hot Flush) and AG-348 Concentration and Relevant AG-348 Pharmacokinetic Parameters
Description: Predicted probability of experiencing all grade hot flush at the doses of 5, 20, and 50 mg mitapivat BID based on exposure-response model.
Time Frame: From first dose of mitapivat to the end of study, including follow-up (up to Day 197)
Population: Safety Set: Participants who were administered the study drug. Participants who received mitapivat in studies: study AG348-C-003 (NCT02476916): 52 participants; study AG348-C-006 (NCT03548220): 40 participants; study AG348-C-007 (NCT03559699): 27 participants; and study AG348-C-011 (NCT03853798): 36 participants, were pooled for the analysis of this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Percent probability
Groups:
- Experimental: AG-348 5 mg: Participants received AG-348 tablets, 5 mg BID, administered orally, for 4 weeks as a starting dose, participants continued to receive the same dose as determined by the investigator based on safety and efficacy up to Week 12, followed by the same optimized dose of 5 mg BID, for a period of 12 weeks as a fixed-dose.
- Experimental: AG-348 20 mg: Participants received AG-348 tablets, starting dose of 5 mg BID for 4 weeks, the dose was uptitrated to 20 mg BID, administered orally, up to Week 12 as an optimized dose as determined by the investigator based on safety and efficacy, followed by the same optimized dose of 20 mg BID further for a period of 12 weeks as a fixed-dose.
- Experimental: AG-348 50 mg: Participants received AG-348 tablets, starting dose of 5 mg BID for 4 weeks, the dose was uptitrated to 20 mg BID, administered orally, up to Week 8 followed by dose up titration to 50 mg BID up to Week 12 as an optimized dose, followed by the same optimized dose of 50 mg BID, as determined by the investigator based on safety and efficacy, further for a period of 12 weeks as a fixed-dose.
Arm/Group | Experimental: AG-348 5 mg | Experimental: AG-348 20 mg | Experimental: AG-348 50 mg
Number analyzed (Participants) | 2 | 3 | 150
Percent probability | 3.37 [1.22 to 7.35] | 4.03 [1.61 to 8.36] | 5.5 [2.48 to 10.5]

17. Other Pre Specified Outcome: Percentage of Participants With Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AESI can be serious or non-serious.
Time Frame: Through 4 weeks after last dose (approximately Week 31)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change From Baseline in Bone Mineral Density Z-Score at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change From Baseline in Bone Mineral Density T-Score at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

20. Secondary Outcome: Exposure-Response Relationship Between Safety Parameters (Sex Hormone in Male Subjects) and AG-348 Concentration and Relevant AG-348 Pharmacokinetic Parameters
Description: Predicted percent change from baseline at Week 24 in the sex hormone measures (total testosterone, free testosterone, and estrone) at the doses of 5, 20, and 50 mg mitapivat BID in male participants.
Time Frame: Baseline, Week 24
Population: Safety Set: Participants who were administered the study drug. Male participants who received mitapivat in studies: study AG348-C-003 (NCT02476916): 32 participants; study AG348-C-006 (NCT03548220):15 participants; study AG348-C-007 (NCT03559699): 7 participants; and study AG348-C-011 (NCT03853798): 14 participants were pooled for analysis of this outcome measure.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Experimental: AG-348 5 mg | Experimental: AG-348 20 mg | Experimental: AG-348 50 mg
Number analyzed (Participants) | 2 | 3 | 63
Percent change
  Total Testosterone | 0.877 [0.41 to 1.43] | 3.18 [1.49 to 5.4] | 7.59 [3.29 to 13.7]
  Free Testosterone | 6.01 [1.66 to 13.2] | 14.1 [4 to 27.5] | 26 [7.14 to 55.1]
  Estrone | -31.5 [-51 to -21.1] | -56.5 [-67.3 to -48.4] | -68.2 [-74.5 to -62.6]

ADVERSE EVENTS:
Time Frame: From time of signing of informed consent form to end of study, including follow-up (up to Day 197)
Description: The placebo arm includes AEs that occurred in participants who received at least 1 dose of AG-348 matching placebo during the study. As pre-specified in SAP, AEs that occurred in AG-348 arms for participants who received AG-348 treatment during the study are reported based on the fixed dose treatment received. The safety analysis set included all participants who received at least 1 dose of study treatment.
Arm/Group | Placebo Comparator: Placebo | Experimental: AG-348, 5 mg | Experimental: AG-348, 20 mg | Experimental: AG-348, 50 mg
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/2 | 0/3 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/39 | 0/2 | 1/3 | 3/35
Other Adverse Events (participants affected / at risk) | 35/39 | 1/2 | 3/3 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator: Placebo (N=39) | Experimental: AG-348, 5 mg (N=2) | Experimental: AG-348, 20 mg (N=3) | Experimental: AG-348, 50 mg (N=35)
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator: Placebo (N=39) | Experimental: AG-348, 5 mg (N=2) | Experimental: AG-348, 20 mg (N=3) | Experimental: AG-348, 50 mg (N=35)
Nausea (Gastrointestinal disorders) | 9 | 0 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 0 | 2 | 3
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 0 | 1 | 4
Influenza like illness (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 13 | 0 | 1 | 5
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 4
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Middle insomnia (Psychiatric disorders) | 3 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2
Initial insomnia (Psychiatric disorders) | 4 | 0 | 0 | 1
Stress (Psychiatric disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of AG-348 and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required

DOCUMENTS (2):
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03548220/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03548220/SAP_002.pdf